CLINICAL TRIAL: NCT03753282
Title: Outcome After Avascular Necrosis of the Femoral Head in Young Patients - Retrospective Analysis With a Min. 10-year Follow-up
Brief Title: Outcome After Avascular Necrosis of the Femoral Head in Young Patients
Acronym: AVN
Status: Withdrawn | Type: Observational
Why Stopped: difficulty enrolling patients, no patient recruited
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-01264; ch18Saxer3
Record Dates: First submitted 2018-11-23; First posted 2018-11-26 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Avascular Necrosis of the Femoral Head
Keywords: Total hip arthroplasty; Total hip replacement
MeSH Terms: conditions — Femur Head Necrosis | interventions — Surveys and Questionnaires; Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Population 1: Patients with a first AVN-related contact (initial or confirmed diagnosis) at the Universitätsspital Basel (USB) or Kantonsspital Basel-Liestal (KSBL) in the years between 1999-2006 (being assessed by questionnaires for patient reported outcome and questionnaire for course of the disease)
  Interventions: Other: questionnaires for patient reported outcome; Other: questionnaire for course of the disease
- Population 2: Patients with a THA because of AVN in the years 2000-2007 (being assessed by questionnaires for patient reported outcome and questionnaire for course of the disease)
  Interventions: Other: questionnaires for patient reported outcome; Other: questionnaire for course of the disease

INTERVENTIONS:
Other: questionnaires for patient reported outcome — questionnaires with respect to outcomes:
  * Reoperations
  * Short term complications
  * Long term complications
  * EQ-5D (current)
  * HOOS (current)
  * disease related change of occupation
  * use of walking aids
  * comorbidities
  * medication
Other: questionnaire for course of the disease — questionnaires to assess course of the disease:
  * from initial diagnosis of AVN to joint replacement as total hip arthroplasty (THA)
  * therapeutic interventions

SUMMARY:
1. The course of AVN between Initial diagnosis and total hip replacement (THA) is analysed. The impact of early interventions versus conservative therapy in AVN before THA will be evaluated.
2. The short and long term outcomes of AVN patients undergoing THA with respect to complications, reoperations and quality of life are investigated. Potential risk factors for adverse outcomes will be investigated.

DETAILED DESCRIPTION:
The study is to describe the course of avascular necrosis (AVN) of the femoral head from initial diagnosis and to collect data on treatment options and the further course in these cases. The duration from initial diagnosis of AVN to joint replacement as total hip arthroplasty (THA) will be analysed and the course after joint replacement with potential short- and long-term complications will be evaluated.

The impact of THA after AVN on activities of daily living will be assessed by Euroquol 5 Dimensions (EQ-5D-5L) and Hip disability and Osteoarthritis Outcome Score (HOOS) questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* MRI of the hip available from diagnosis at the USB or KSBL Liestal
* Informed Consent

Exclusion Criteria:

* Insufficient knowledge of project languages (English, German, French)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Population 1: Patients with a first AVN-related contact (initial or confirmed diagnosis) at the USB or KSBL Liestal in the years between 1999-2006.
  Population 2: Patients with a THA because of AVN at the USB or KSBL Liestal in the years 2000-2007.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-03-05 (Actual)

PRIMARY OUTCOMES:
arthroplasty-free interval (time until THA) | single time point assessment at baseline
  time from first diagnosis of AVN to joint replacement = time to event data (in the years between 1999-2006)
rate of reoperations after THA | single time point assessment at baseline
  reoperation after THA = time to event data (in the years between 2000-2007)

SECONDARY OUTCOMES:
Hip disability and Osteoarthritis Outcome Score (HOOS) | single time point assessment at baseline
  40 item questionnaire to assess patient-relevant outcomes in five separate subscales (pain, symptoms, activity of daily living, sport and recreation function and hip related quality of life). Scores are: None, Mild, Moderate, Severe, Extreme
Euroquol 5 Dimensions (EQ-5D-5L) | single time point assessment at baseline
  Five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.

CONTACTS AND LOCATIONS:
Overall Officials: Franziska Saxer, Dr. med, Principal Investigator — Dep. of Orthopedic and Trauma Surgery; University Hospital Basel